CLINICAL TRIAL: NCT06155682
Title: Cognitive and Neural Correlates of TMS Motor Intracortical Inhibition in Schizophrenia
Brief Title: TMS for Inhibition Enhancement in Schizophrenia
Acronym: TIES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephanie Hare, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HP-00108871
Record Dates: First submitted 2023-11-22; First posted 2023-12-04 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
Keywords: TMS; brain inhibition; SICI; schizophrenia; fMRI
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): multiple trains of active transcranial magnetic stimulation in a day (using the active TMS coil), for multiple days
  Interventions: Device: repetitive transcranial magnetic stimulation (active)
- sham rTMS (Sham Comparator): multiple trains of sham transcranial magnetic stimulation in a day (using the sham comparator TMS coil), for multiple days
  Interventions: Device: repetitive transcranial magnetic stimulation (sham)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (active) — non-invasive active repetitive stimulation applied to the scalp surface
  Arms: Active rTMS
Device: repetitive transcranial magnetic stimulation (sham) — non-invasive active repetitive stimulation applied to the scalp surface
  Arms: sham rTMS

SUMMARY:
This study purpose is to perform a pilot mechanistic trial repetitive transcranial magnetic stimulation (rTMS) clinical trial in 34 people with schizophrenia (Sz). The trial will evaluate whether inhibitory 1 Hertz (Hz) rTMS targeting motor cortex can increase brain inhibition reflected in a decrease in the short-interval intracortical inhibition (SICI) score from pre-to-post-treatment. We will also collect preliminary data on the effect of rTMS on the resting functional connectivity of the motor cortex and other brain regions and the relationship of change in SICI to change in cognitive performance

DETAILED DESCRIPTION:
This study is a randomized double blind clinical trial being funded by the National Institute of Mental Health (NIMH). The primary aim is to estimate feasibility and tolerability of a 5-day, 1Hz rTMS intervention in 34 participants with schizophrenia. A secondary aim is to assess target engagement by investigating whether 1 Hz rTMS applied to motor cortex can enhance intracortical inhibition in participants with schizophrenia. The participants with Sz will be randomized in a 1:1 ratio to either active 1Hz rTMS or sham 1Hz rTMS. We do not necessarily anticipate a statistically significant difference between treatment groups, given our limited sample size. Rather, we are focused on generating effect size estimates that will help us determine whether and how to proceed to the next phase of research and a future R01 submission. We will explore the relationship between change in SICI score (pre-to-post-treatment) and total scores of clinical scales (Fagerstrom nicotine dependence, the brief psychiatric rating scale and the brief negative symptoms scale) and medication dose and type. We will also collect preliminary data on the effect of rTMS on the resting state functional connectivity of the motor cortex with other brain regions, and the change performance on cognitive tasks (i.e., stop signal reaction time, spatial working memory) from pre-to-post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years
2. Male or Female
3. Able to participate in the informed consent process and provide voluntary informed consent.
4. A Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) diagnosis of schizophrenia documented by the Structured Clinical Interview for DSM-5 (SCID-5)

Exclusion Criteria:

1. A history of a DSM-5 substance misuse disorder (other than caffeine or tobacco or mild marijuana misuse) within the past six months; or a positive baseline urine drug screen.
2. A history of a current neurological disorder (including, but not limited to Parkinson's Disease, epilepsy, or Multiple Sclerosis)
3. History of head trauma resulting in unconsciousness
4. Contraindications for TMS, including any history of seizure other than febrile seizure, presence of ferromagnetic metal in cranium, presence of cochlear implant, presence of deep brain stimulation (DBS) electrodes based on medical history
5. Contraindications for MRI, including pacemakers or other metal in body
6. Suspected DSM-5 intellectual disability based upon clinical interview and psychosocial history
7. Pregnancy
8. Any change in type of antipsychotic medication in the last 30 days and dose in the last 14 days
9. Treatment with a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or greater or any anticonvulsant due to the potential of these medications to affect TMS SICI score and the efficacy of rTMS
10. Prior history of rTMS treatment in the past 5 years
11. Endorsement of active suicidal ideation on the Columbia-Suicide Severity Rating Scale (version: last 30 days) reflected by "yes" response on items 3, 4, or 5 of the ideation questions and/or "yes" to any of the four suicidal behavior items (actual attempt, interrupted attempt, aborted attempt, preparatory acts/behavior)
12. A score of 7 or more on the Simpson-Angus Scale of Extrapyramidal Symptoms (range 0-52 with higher scores indicating worse extrapyramidal symptoms)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
The change in the short interval intracortical inhibition (SICI) score | one week
  At baseline, and at the end of 5 days of rTMS treatment, we will perform 24 trials of paired-pulse TMS to calculate SICI score (defined as the ratio of the evoked motor potential to the paired-pulse TMS in our SICI protocol relative to a single suprathreshold pulse). We will average across these 24 trials to get an average SICI score (both pre-TMS and post-TMS). We will calculate the change in SICI score (pre-TMS to post-TMS) for each participant.

SECONDARY OUTCOMES:
change in motor cortex functional connectivity | one week
  The measure will be collected at baseline (pre-treatment) and after week 1 (post-treatment). At each magnetic resonance imaging (MRI) scanning session, we will conduct a resting functional MRI scan. The mean of motor functional connectivity will be defined as the average connectivity between regions of interest in the motor network that is informed by our preliminary data and Research Aim 2. We will use the pre- and post- rTMS functional connectivity values to calculate change in motor functional connectivity.
change in neurocognitive performance | one week
  This measure will be collected at baseline (pre-treatment) and after week 1 (post-treatment). We will also collect preliminary data on the effect of rTMS on the relationship of change in SICI to change in neurocognitive performance. Neurocognitive data will include Stop-Signal task performance, working memory performance, and total and subscale scores on the the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery (MCCB). We will use the pre- and post- rTMS neurocognitive scores to calculate change in neurocognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Hare, PhD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu